CLINICAL TRIAL: NCT02149212
Title: Randomized Double-blind Trial Between Clinical and Endovascular Treatment in Patients With Advanced Chronic Venous Insufficiency and Iliac Venous Obstruction
Brief Title: Iliac Vein Stenting in Advanced Chronic Venous Insufficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Fabio H Rossi, PHD, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDPC_2 2014
Record Dates: First submitted 2014-05-25; First posted 2014-05-29 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Iliac Vein Obstruction; May-Thurner Syndrome; Cockett Syndrome
Keywords: Iliac; Vein; Stent
MeSH Terms: conditions — May-Thurner Syndrome | interventions — aminaftone; Stents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinical Treatment (Active Comparator): Phlebotonics: Aminaftone 75 mg BID Limb elastic compression support (Elastic stockings: Venosan / Elastic Bandages: Atamed) Unna boot dressing
  Interventions: Drug: Phlebotonic; Procedure: Limb elastic compression support; Procedure: Unna boot dressing
- Iliac vein stenting (Active Comparator): Wallstent
  Interventions: Drug: Phlebotonic; Device: Stent; Procedure: Limb elastic compression support; Procedure: Unna boot dressing

INTERVENTIONS:
Drug: Phlebotonic — Aminaftone -- 75 mg BID
  Other Names: Aminaftone
Device: Stent — Iliac Vein Stenting
  Other Names: Wallstent
  Arms: Iliac vein stenting
Procedure: Limb elastic compression support — CEAP 3-5 > 20-30 mmHg compression stockings CEAP 6 > elastic bandages
  Other Names: Venosan compression stockings; Atamed elastic bandages
Procedure: Unna boot dressing — CEAP 6 > Unna boot dressing

SUMMARY:
About 90 % of vascular symptoms affecting the lower limbs consist of venous diseases. Its highest incidence occurs from the second decade of life, affecting significantly the economically active population. Chronic Venous Insufficiency treatment aims to relieve symptoms, treat and prevent complications, prevent recurrences and provide cosmetic satisfaction with minimal side effects. It's current treatment includes some classic postural measures (leg elevation), elastic stockings and bandages compression therapy and possible medication (phlebotonics). The results in the medium and long term are unfavorable, since a large number of patients do not get better or evolves with recurrence of symptoms. Nowadays many, no prospective , not randomized , international studies have shown favorable results with endovascular treatment of obstruction in the iliac vein territory in patients with advanced Chronic Venous Insufficiency . The purpose of this prospective, double-blinded randomized study is to evaluate the results obtained with endovascular treatment, through the use of angioplasty and stenting in this group of patients when compared with clinical treatment .

ELIGIBILITY:
Inclusion Criteria:

* Advanced Chronic Venous Insufficiency (CEAP 3-6) submitted to clinical treatment for at least 1 year with no response.
* Subject must be > 18 and < 80 years of age
* Willing to participate in and able to understand, read and sign the informed consent document before the planned procedure
* On duplex ultrasound: patent common femoral vein, and patent deep femoral vein, and/or femoral vein of the study leg

Exclusion Criteria:

* Subject cannot or will not provide written informed consent
* Previous venous stent implantation involving the study leg or inferior vena cava
* Previous venovenous bypass surgery involving the study leg
* Known metal allergy precluding endovascular stent implantation
* Known reaction or sensitivity to iodinated contrast that cannot be managed with premedication
* Subjects who are pregnant (women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment
* Acute deep venous thrombosis involving either leg
* Known history of chronic total occlusion of the common femoral vein of the study leg.
* Known history of thrombophilia (e.g., protein C or S deficiency, anti-thrombin III deficiency, presence of lupus anticoagulant, etc.)
* Venous compression caused by tumor encasement
* Venous outflow obstruction caused by tumor thrombus
* Life expectancy of less than 6 months
* Lower Extremity Arterial Insufficiency
* Elevated baseline blood creatinine (value greater than the upper limit of the normal range)
* Any concurrent disease or condition that, in the opinion of the Investigator, would make the subject unsuitable for participation in the study; examples include but are not limited to the inability to lie supine for the index procedure (e.g., severe congestive heart failure), thrombocytopenia or other hematological disorders associated with an unacceptable risk of bleeding, implanted orthopedic hardware that precludes proper imaging, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on the Pain Visual Analogue Sacale at 6 months | 6 months
Venous ulcer cicatrization at 6 months | 6 months

SECONDARY OUTCOMES:
Change from the baseline Venous Clinical Severity Score at 6 month | 6 months
Change from baseline in SF-36 Quality of Life questionnaire at 6 months | 6 months
Stent integrity at 6 months | 6 months
Stent position at 6 months | 6 months
  Pelvic X-ray
Stent patency at 6 months | 6 months
  Stent patency obtained with treated venous segment Duplex Scanning

CONTACTS AND LOCATIONS:
Overall Officials: Fabio H Rossi, PHD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (1):
- Instituto Dante Pazzanese de Cardilogia, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Alhalbouni S, Hingorani A, Shiferson A, Gopal K, Jung D, Novak D, Marks N, Ascher E. Iliac-femoral venous stenting for lower extremity venous stasis symptoms. Ann Vasc Surg. 2012 Feb;26(2):185-9. doi: 10.1016/j.avsg.2011.05.033. Epub 2011 Oct 22. PMID 22018502
- [Background] Kolbel T, Lindh M, Akesson M, Wasselius J, Gottsater A, Ivancev K. Chronic iliac vein occlusion: midterm results of endovascular recanalization. J Endovasc Ther. 2009 Aug;16(4):483-91. doi: 10.1583/09-2719.1. PMID 19702343
- [Background] Raju S. Best management options for chronic iliac vein stenosis and occlusion. J Vasc Surg. 2013 Apr;57(4):1163-9. doi: 10.1016/j.jvs.2012.11.084. Epub 2013 Feb 20. PMID 23433816
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829
- [Derived] Lorencao de Almeida B, Rossi FH, Guerra de Moraes Rego Sousa A, Kambara AM, Izukawa NM, Beteli CB, Andrade Cavalcante SF, Rodrigues TO, Thorpe PE. Correlation between venous pressure gradients and intravascular ultrasound in the diagnosis of iliac vein compression syndrome. J Vasc Surg Venous Lymphat Disord. 2018 Jul;6(4):492-499. doi: 10.1016/j.jvsv.2017.11.015. Epub 2018 Mar 8. PMID 29526687
- [Derived] Rossi FH, Kambara AM, Izukawa NM, Rodrigues TO, Rossi CB, Sousa AG, Metzger PB, Thorpe PE. Randomized double-blinded study comparing medical treatment versus iliac vein stenting in chronic venous disease. J Vasc Surg Venous Lymphat Disord. 2018 Mar;6(2):183-191. doi: 10.1016/j.jvsv.2017.11.003. Epub 2017 Dec 29. PMID 29292114